CLINICAL TRIAL: NCT02528734
Title: Impact of Pneumothorax Duration Before Treatment on the Success of Needle Exsufflation
Brief Title: Prospective Evaluation of Needle Exsufflation for Pneumothorax
Status: Completed | Type: Observational
Sponsor: Hôpital Louis Mourier (Other)
Responsible Party: Principal Investigator, Prof Jean-Damien RICARD, Professor in Intensive Care Medicine, Assistant Head of Medico-Surgical ICU, Hôpital Louis Mourier
Other Study IDs: HLM_JDR5
Record Dates: First submitted 2015-08-17; First posted 2015-08-19 (Estimated); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: Pneumothorax
Keywords: pneumothorax
MeSH Terms: conditions — Pneumothorax

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Monocentric observational study of needle exsufflation for pneumothorax in the ICU.

DETAILED DESCRIPTION:
The main objective of this prospective observational non interventional study is to investigate a possible relationship between prior duration of pneumothorax (defined as the duration from first occurence of chest pain reported by patient to exsufflation) and the success of exsufflation procedure (defined by the absence of a chest tube insertion in the following 24h).

ELIGIBILITY:
Inclusion Criteria:

* adult ICU patients requiring needle exsufflation for spontaneous pneumothorax

Exclusion Criteria:

* refuse to participate
* contraindications to needle exsufflation (acute respiratory failure requiring immediate chest tube insertion)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients admitted to the ICU with a pneumothorax
Sampling Method: Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Number of patients with early success of needle exsufflation | 24 hrs
  success of needle exsufflation is defined as the absence of chest tube insertion requirement within 24hrs following needle exsufflation
Number of patients with early success of needle exsufflation with duration of symptoms prior to exsufflation greater than 48 hrs | 24 hrs
  success of needle exsufflation is defined as the absence of chest tube insertion requirement within 24hrs following needle exsufflation; duration of symptoms prior to exsufflation is the time (in hrs) elapsed between first chest pain reported by the patient and needle exsufflation

SECONDARY OUTCOMES:
Length of ICU stay | 8 days
  participants will be followed for the duration of ICU stay, from ICU admission to ICU discharge, an expected average of 8 days
Length of hospital stay | 15 days
  participants will be followed for the duration of hospital stay, from hospital admission to hospital discharge, an expected average of 15 days
Number of patients requiring early surgical pleurodesis because of persistent pneumothorax | 8 days
  Patients will be monitored for eventual need for surgical pleurodesis during their ICU stay because of persistent or worsening pneumothorax
Number of patients with late exsufflation failure | 8 days
  late exsufflation failure is defined as patients requiring chest tube insertion at least 24 hrs after needle exsufflation because of persistent or worsening of pneumothorax despite initial early success

OTHER OUTCOMES:
Number of patients with pneumothorax recurrence | 30 days
  Patients will be followed for an expected average of 30 days to identify those with recurrent pneumothorax
Maximal patient self-reported pain during procedure | 30 mintutes
  patients are asked to assess the maximal pain felt during needle exsufflation or chest tube insertion with the use of a numeric scale from 0 [no pain] to 10 [worst possible pain]
Number of patients with treatment-related adverse event | 8 days
  Patients will be followed for 8 days to identify those with either hemothorax (defined as hematic pleural effusion requiring thoracic drainage); or a vacuo pulmonary edema (defined as occurrence of localised alveolar interstitial opacities on post-procedure chest X-ray); or site of chest tube insertion infection (presence of purulent secretions issuing from chest tube insertion site)

CONTACTS AND LOCATIONS:
Overall Officials: Ricard Jean-Damien, MD, PhD, Study Director — Hopital Louis Mourier
Locations (1):
- Louis Mourier Hospital, Colombes, France

REFERENCES:
- [Background] MacDuff A, Arnold A, Harvey J; BTS Pleural Disease Guideline Group. Management of spontaneous pneumothorax: British Thoracic Society Pleural Disease Guideline 2010. Thorax. 2010 Aug;65 Suppl 2:ii18-31. doi: 10.1136/thx.2010.136986. No abstract available. PMID 20696690
- [Result] Andrivet P, Djedaini K, Teboul JL, Brochard L, Dreyfuss D. Spontaneous pneumothorax. Comparison of thoracic drainage vs immediate or delayed needle aspiration. Chest. 1995 Aug;108(2):335-9. doi: 10.1378/chest.108.2.335. PMID 7634863
- [Derived] Vuillard C, Dib F, Achamlal J, Gaudry S, Roux D, Chemouny M, Javaud N, Dreyfuss D, Ricard JD, Messika J. Longer symptom onset to aspiration time predicts success of needle aspiration in primary spontaneous pneumothorax. Thorax. 2019 Aug;74(8):780-786. doi: 10.1136/thoraxjnl-2019-213168. Epub 2019 Jun 12. PMID 31189731